CLINICAL TRIAL: NCT03736408
Title: Frequency of Occurrence of the Pain Form of Temporomandibular Joint Dysfunction
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Malgorzata Pihut, Head of Department of Prosthetic Dentistry, Clinical Professor, Jagiellonian University
Other Study IDs: 1072.6120.57.2018
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Temporomandibular Disorders
Keywords: temporomandibular joint dysfunction; pain form; treatment; epidemiologcal assessment
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. Group without Pain - TMJ disorders symptoms: 1. The symptoms concerning joints were: the type of sound symptoms (clicking or popping), their frequency and the phase of the movement of lowering and lifting the jaw during which they occurred, occurrence of the tension type headache or back pain. Hypertension of the mastication muscles is frequently connected with a parafunction activity like grinding or clenching the teeth, which cause abnormal pressure on the joints
- 2. Group with Pain and symptoms TMJ disorder: The pain form of the disease is manifested by spontaneous pain in the preaural region, accompanied by pain or tenderness of the mastication muscle. Pain that appears during palpation examination of temporomandibular joints is frequently not related to inflammation of the soft tissue around the temporomandibular joints, as it is claimed by several authors of the paper. The cause of this problem is a long-term overload of soft tissue causally associated with excessive muscle tension, that sometimes even persists for years

SUMMARY:
Temporomandibular joint dysfunction (TMJD) includes disorders of the masticatory muscles in the stomatognathic system, temporomandibular joints and the surrounding structures. They are often associated with abnormal conditions of occlusion. The term "functional disorders" does not include all diseases of the muscular and joint system, like inflammatory, degenerative changes and cancer lesions of the muscles (multiple sclerosis, tetany, dermatomyositis). They are often the result of excessive and prolonged muscle hyperactivities and excessive work that cause non-physiological loads occurring in temporomandibular joints

DETAILED DESCRIPTION:
Temporomandibular joint dysfunction (TMJD) includes disorders of the masticatory muscles in the stomatognathic system, temporomandibular joints and the surrounding structures. They are often associated with abnormal conditions of occlusion. The term "functional disorders" does not include all diseases of the muscular and joint system, like inflammatory, degenerative changes and cancer lesions of the muscles (multiple sclerosis, tetany, dermatomyositis). They are often the result of excessive and prolonged muscle hyperactivities and excessive work that cause non-physiological loads occurring in temporomandibular joints.

Certainly the most common complaint in this group of patients is muscle pain, which may range from slight tenderness to extreme discomfort. However, the origin of that pain is most often associated with increased levels of muscular use. Clinically this is seen as an inability to open the mouth widely. The restriction may be at any degree of opening depending on where the discomfort is felt. Local muscle soreness is a primary non-inflammatory muscular pain discomfort. It is often the first response of the muscle tissue to prolonged excessive contraction and is the most common type of acute muscle pain in dental practice.

The pain form of the disease is manifested by spontaneous pain in the preaural region, accompanied by pain or tenderness of the mastication muscle. Pain that appears during palpation examination of temporomandibular joints is frequently not related to inflammation of the soft tissue around the temporomandibular joints, as it is claimed by several authors of the paper. The cause of this problem is a long-term overload of soft tissue causally associated with excessive muscle tension, that sometimes even persists for years.

Due to an etiological factor, very important information associated with emotional tension and stress as well as sleep disturbances in relation to other pain complaints were verified.

The aim of the study was to carry out a retrospective assessment of the frequency of the pain form of functional disorders based on the analysis of medical records (results of a physical examination and a specialized functional test) of patients treated at the Consulting Room of Temporomandibular Joint Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* pain and painless form of temporomandibular joints dysfunction,
* required age range (>18 years)
* good general state of health

Exclusion Criteria:

* the will of the patient,
* emergence of general diseases,
* trauma,
* local inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study enrolled a group of 334 patients of both sexes, who reported to the prosthodontic treatment in Consulting Room of Temporomandibular Joint Dysfunction at Dental Institute at Jagiellonian University in Cracow, between January 2015 to June 2018, due to the pain and painless form of the temporomandibular joints dysfunctions.
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison of pain and painless type of the temporomandibular joint disorders. | 12 months
  The aim of the study was to carry out a retrospective assessment of the frequency of the pain form of functional disorders based on the analysis of medical records (results of a physical examination and a specialized functional test) of patients treated at the Consulting Room of Temporomandibular Joint Dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Pihut, Prof., Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian University Department of Prosthetic Dentistry, Krakow, Lesser Poland Voivodeship, Poland